CLINICAL TRIAL: NCT04782115
Title: Protein by Dual Blockage of VEGF and FGF-2) in Subjects With Diabetic Macular Edema.
Brief Title: Evaluation of RC28-E Injection in Diabetic Macular Edema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 28C002
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — KH902 fusion protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 1.0mg RC28-E injection Q8 (Experimental): In the loading phase (from week 0 to week 8), the study eye will receive intravitreal injection of 1.0 mg RC28-E every 4 weeks, for 3 consecutive times; From then on to the 48th week, the patients were visited every 4 weeks and given medicine every 8 weeks.
  Interventions: Biological: intravitreal injection of RC28-E
- 1.0mg RC28-E injection as needed (Experimental): In the loading phase (from week 0 to week 16), the study eye will receive intravitreal injection of 1.0mg RC28-E every 4 weeks, for 5 consecutive times;In the as needed (pro re nata,PRN)phase (from then on to week 48), the study eye will receive the same dose on an PRN schedule based upon the physician assessment in accordance with pre-specified criteria.
  Interventions: Biological: intravitreal injection of RC28-E
- 2.0mg RC28-E injection Q8 (Experimental): In the loading phase (from week 0 to week 8), the study eye will receive intravitreal injection of 2.0mg RC28-E every 4 weeks, for 3 consecutive times; From then on to the 48th week, the patients were visited every 4 weeks and given medicine every 8 weeks.
  Interventions: Biological: intravitreal injection of RC28-E
- 2.0mg RC28-E injection as needed (Experimental): In the loading phase (from week 0 to week 16), the study eye will receive intravitreal injection of 2.0mg RC28-E every 4 weeks, for 5 consecutive times;In the as needed (pro re nata,PRN)phase (from then on to week 48), the study eye will receive the same dose on an PRN schedule based upon the physician assessment in accordance with pre-specified criteria.
  Interventions: Biological: intravitreal injection of RC28-E
- control group (Experimental): In the loading phase (from week 0 to week 8), the study eye will receive intravitreal injection of Conbercept every 4 weeks, for 3 consecutive times;In the as needed (pro re nata,PRN)phase (from then on to week 48), the study eye will receive the same dose on an PRN schedule based upon the physician assessment in accordance with pre-specified criteria.
  Interventions: Biological: Conbercept

INTERVENTIONS:
Biological: intravitreal injection of RC28-E — a chimric decoy receptor trap fusion protein by dual blockage of VEGF and FGF
  Arms: 1.0mg RC28-E injection Q8; 1.0mg RC28-E injection as needed; 2.0mg RC28-E injection Q8; 2.0mg RC28-E injection as needed
Biological: Conbercept — KH902(Conbercept）
  Arms: control group

SUMMARY:
This is a non-randomized, open-label, multicenter, 48-week study to investigate the efficacy, safety and pharmacokinetics of RC28-E injection in the treatment of patients with diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

* Sign the consent form, willing and able to comply with clinic visits and study-related procedures;
* Aged 18 years to 80 years, male or female;
* Diabetes mellitus(type 1 or 2);
* The study eye must followed:

  1. Retinal thickening secondary to diabetes mellitus (DME) involving the center of the fovea; Decrease in vision determined to be primarily the result of DME and not to other causes.
  2. BCVA score in the study eye of 73 to 24 using the ETDRS protocol at an initial testing distance of 4 meters.
  3. The central subfield thickness ≥300μm in the center subfield as assessed on OCT by the reading center;
* If both eyes meet the inclusion criterion, one eye with poor BCVA is selected as the study eye; the researchers judged that the fellow eye should not be treated with other anti-VEGF drugs recently.

Exclusion Criteria:

* The macular edema caused by others instead of diabetes mellitus;
* Structural damage to the center of the macula in the study eye that is likely to preclude improvement in BCVA following the resolution of macular edema including atrophy of the retinal pigment epithelium, subretinal fibrosis or scar, significant macular ischemia or organized hard exudates;
* Current iris neovascularization, vitreous hemorrhage, tractional retinal detachment or epiretinal membrane involving the macula in the study eye;
* Only one functional eye even if that eye is otherwise eligible for the study;
* Evidence of periocular or intraocular inflammation or infection including infectious blepharitis, keratitis, scleritis, conjunctivitis, endophthalmitis or uveitis at screening assessment in either eye;
* Previous treatment with anti-angiogenic drugs in either eye or system (ranibizumab, aflibercept, conbercept, etc) within 3 months of the Day 0;
* History of cardiovascular and cerebrovascular events within 6 months of screening visit: myocardial infarction, unstable angina pectoris, ventricular arrhythmias, New York heart association grade II + heart failure, stroke, etc.;
* Uncontrolled clinical disease (such as severe psychiatric, neurological, cardiovascular, respiratory disease or other systemic diseases) and tumors;
* Those who participated in clinical trials for 3 months or 5 half-lives of the investigational product (the longer the time) before the baseline period;
* Those who considered unsuitable for enrollment by investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in BCVA at 24 week; | Baseline,week 24
  BCVA=Best-corrected visual acuity;Measurement of visual acuity with Early Treatment Diabetic Retinopathy Study (ETDRS) charts.
Mean change from baseline in BCVA at 52 week; | Baseline, Week 52
  Measurement of visual acuity with Early Treatment Diabetic Retinopathy Study (ETDRS) charts.

SECONDARY OUTCOMES:
Mean change from baseline in BCVA at every visit during treatment period; | Baseline up to Week 52
  Measurement of visual acuity with Early Treatment Diabetic Retinopathy Study (ETDRS) charts.
Mean change from baseline in central subfield thickness at 12, 24, 36, 52 week. | 12, 24, 36, 52 week.
  Measurement of central subfield thickness by OCT.
Percentage of subjects with VA improvement (who gained >0 letters, ≥5 letters, ≥10 letters, ≥ 15 letters in their BCVA) from baseline at 52 week; | Baseline up to Week 52
  Measurement of visual acuity with Early Treatment Diabetic Retinopathy Study (ETDRS) charts.
Percentage of subjects with VA worsen (who lost ≥5 letters, ≥10 letters, ≥15 letters in their BCVA) from baseline at 52 week; | Baseline, Week 52
  Measurement of visual acuity with Early Treatment Diabetic Retinopathy Study (ETDRS) charts.
Percentage of subjects with BCVA ≥ 68 letters(a visual acuity Snellen equivalent of 20/40 or better) at 52 week; | Baseline, Week 52
  Measurement of visual acuity with Early Treatment Diabetic Retinopathy Study (ETDRS) charts.
Frequency of administration RC28-E; | Baseline, Week 52
  Number of intravitreal injections
Safety of RC28-E injection | Baseline up to Week 52
  Incidence of AE in ocular and non-ocular

CONTACTS AND LOCATIONS:
Locations (37):
- China (37):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Aier Intech Eye Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Zhongshan Ophthalmic Center of Sun Yat-sen University, Guangzhou, Guangdong
  - Huizhou Central People's Hospital, Huizhou, Guangdong
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The First People's Hospital of Zunyi, Zunyi, Guizhou
  - CNPC Central Hospital, Langfang, Hebei
  - Hebei Eye Hospital, Xingtai, Hebei
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan Provincial Eye Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Zhengzhou Second Hospital, Zhengzhou, Henan
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - The Affiliated Eye Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The Affiliated Eye Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Shenyang He Eye Specialist Hospital, Shenyang, Liaoning
  - The Fourth People's Hospital of Shenyang, Shenyang, Liaoning
  - People's Hospital of Ningxia Hui Autonomous Region, Yinchuan, Ningxia
  - Weifang Eye Hospital, Weifang, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Shanxi Eye Hospital, Taiyuan, Shanxi
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Ruian People's Hospital, Rui’an, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang W, Cheng S, Gu X, Liu X, Dai H, Zhuang W, Sun B, Gao L, Sun X, Zhang M, Song Z, Wang W, Li L, Chen H, Fang J, Chen Y. Simultaneous inhibition of fibroblast growth factor-2 and vascular endothelial growth factor-a with RC28-E in diabetic macular edema: a phase 2 randomised trial. Br J Ophthalmol. 2025 Jun 23;109(7):784-790. doi: 10.1136/bjo-2024-326006. PMID 40122579